CLINICAL TRIAL: NCT00297544
Title: Effect of Sildenafil on Endothelial Function
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rambam Health Care Campus (Other)
Collaborators: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Educational/Counseling/Training
Other Study IDs: 1777-CTIL
Record Dates: First submitted 2006-02-27; First posted 2006-02-28 (Estimated); Last update posted 2006-02-28 (Estimated); Status verified 2005-11

CONDITIONS: Impotence
Keywords: impotence; endothelial function; autonomic nervous system
MeSH Terms: conditions — Erectile Dysfunction | interventions — Sildenafil Citrate

INTERVENTIONS:
Drug: Viagra

SUMMARY:
We are investigating the chronic effect of daily assumption of Viagra on the blood vessels function in patients with impotence. The study will include 2 groups: 1- patients with multiple risk factors, e.g. hypertension 2- patients with no cardiovascular risk factors

DETAILED DESCRIPTION:
We are investigating the chronic effect of daily assumption of Viagra on the blood vessels function in patients with impotence. The study will include 2 groups: 1- patients with multiple risk factors, e.g. hypertension 2- patients with no cardiovascular risk factors

ELIGIBILITY:
Inclusion Criteria:

* age 40-70
* impotence
* with and without hypertension, Hypercholesteremia or DM

Exclusion Criteria:

* CHF: NYHA > II
* Stable angina: CCS > II
* Nitrate treatment

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2005-10

PRIMARY OUTCOMES:
Improvement of endothelial function following Viagra treatment, according to platismographia.

CONTACTS AND LOCATIONS:
Overall Officials: Giris Jacob, Prof, MD, DSc, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Medical Center, Recanati Autonomic Dysfunction CTR, Haifa, Israel

REFERENCES:
- [Background] Dayan L, Greunwald I, Vardi Y, Jacob G. A new clinical method for the assessment of penile endothelial function using the flow mediated dilation with plethysmography technique. J Urol. 2005 Apr;173(4):1268-72. doi: 10.1097/01.ju.0000152290.71948.bf. PMID 15758774
- [Derived] Vardi Y, Appel B, Ofer Y, Greunwald I, Dayan L, Jacob G. Effect of chronic sildenafil treatment on penile endothelial function: a randomized, double-blind, placebo controlled study. J Urol. 2009 Dec;182(6):2850-5. doi: 10.1016/j.juro.2009.08.025. Epub 2009 Oct 17. PMID 19837434